CLINICAL TRIAL: NCT05025527
Title: Biparametric MRI in Prostate Cancer Screening: a Noninferior Randomized Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2021076
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; screen; bpMRI; PSA
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bpMRI (Experimental): Man receive the bpMRI for Prostate cancer(PCa) screening
  Interventions: Diagnostic Test: biparametric MRI (bpMRI)
- PSA (Active Comparator): Man receive the PSA blood test for Prostate cancer screening
  Interventions: Diagnostic Test: Prostate cancer antigen (PSA)

INTERVENTIONS:
Diagnostic Test: biparametric MRI (bpMRI) — Men go for the bpMRI for PCa (prostate cancer) screening, those who had a suspicious result will go for the next confirmation test
  Arms: bpMRI
Diagnostic Test: Prostate cancer antigen (PSA) — Men go for the PSA test for PCa screening, those who had a suspicious result will go for the next confirmation test
  Arms: PSA

SUMMARY:
This is a single centre non-inferiority randomized controlled trial in comparison of the bpMRI between the traditional pathway in prostate cancer screening

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 80 years old
2. life-expectancy at least 10 years
3. fully understand the clinical trial protocol and sign the informed consent;

Exclusion Criteria:

1. Already diagnosis with prostate cancer;
2. cannot tolerate prostate biopsy or has contraindication to biopsy;
3. cannot tolerate prostate biopsy or has contraindication to MRI examination;
4. undergo biopsy within 1 year
5. patients judged by the investigator to be unsuitable to participate in the clinical trial;

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of men with clinically significant cancer | Within 1 month after the biopsy
  The presence of a single biopsy core indicating disease of ISUP( international society of urological pathology) 2 or more

SECONDARY OUTCOMES:
The proportion of men with clinically insignificant cancer | Within 1 month after the biopsy
  The presence of a single biopsy core indicating disease of ISUP( international society of urological pathology) 1
The proportion of men who do not undergo biopsy | Within 1 month after the biopsy
  The proportion of men who do not need for further biopsy in this trial
The proportion of men with adverse events after the intervention | Within 1 week after the biopsy
  Any of the adverse events during the trial

CONTACTS AND LOCATIONS:
Overall Officials: Haifeng Wang, Principal Investigator — Shanghai East Hospital,Tongji University School of Medicine
Locations (1):
- Shanghai East Hospital, Tongji University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Once available, the results of this trial will be disseminated to an international peer-reviewed journal and presentations at international or national academic conferences. The data will be made available upon request to researchers a) who provide a methodologically sound proposal and b) whose proposed use of the data has been approved by an independent ethical review committee
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available after publication with no end date